CLINICAL TRIAL: NCT00368784
Title: T Cell Repertoire Analysis of Immune Mediated Skin Diseases
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 335144
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2021-03

CONDITIONS: Psoriasis; Mycosis Fungoides
MeSH Terms: conditions — Psoriasis; Mycosis Fungoides

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fifteen tablespoons of blood will be collected prior to the initiation of a treatment and again after the patient shows a clinical response to a treatment. The time between blood draws will be no less than 3 months. There will be no more than two blood draws per patient.
  Blood samples will be used to determine the patient's HLA haplotype via PCR and DNA sequencing. After the patient's haplotype has been established the activated T cell repertoire will be analyzed for clonal expansions. Clonal expansions in the T cell repertoire will be determined by immunoscope analysis, which is a PCR based technique.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Individuals ages 12-85 with an immune mediated skin disease, such as psoriasis, scleroderma, or mycosis fungoides. Peripheral blood and/or check swabs will be collected from participants ages 12- 85 years old. These samples will then be used to characterize the inflammatory cells as described above.
- 2: Age-Matched Controls without immune mediated skin diseases. Peripheral blood and/or check swabs will be collected from participants ages 12- 85 years old. These samples will then be used to characterize the inflammatory cells as described above.

SUMMARY:
This study is designed to identify the cells of the immune system that cause skin disease such as psoriasis and mycosis fungoides. Blood samples from many patients will be compared in hopes of finding common cells and molecules responsible for skin diseases. Results of this study will increase our knowledge about immune mediated skin disease.

DETAILED DESCRIPTION:
The aim of the study is to characterized the T cell repertoire of individuals with immune mediated skin disease (e.g. psoriasis and mycosis fungoides). Peripheral blood with be collected from volunteers with psoriasis, mycosis fungoides and age matched controls. Fifteen tablespoons of blood will be collected prior to the initiation of treatment and again after the patient shows a clinical response to treatment. The time between blood draws will be no less than 3 months. There will be no more than two blood draws per patient. Blood samples will be used to determine the patient's HLA haplotype via PCR and DNA sequencing. After the patient's haplotype has been established the activated T cell repertoire will be analyzed for clonal expansions. Clonal expansions in the T cell repertoire will be determined by immunoscope analysis, which is a PCR based technique.

ELIGIBILITY:
Inclusion Criteria:

* Have an immune mediated skin disease, such as psoriasis or mycosis fungoides
* Are not taking immunosuppressive medications, which may interfere with T cell analysis.

Exclusion Criteria:

* are taking immunosuppressive medications, which may interfere with T cell analysis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects aged 18 years to 55 years who have an immune mediated skin disease, such as psoriasis or mycosis fungoides, and age-matched controls (subjects who do not have an immunce midiated skin disease).
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2007-01; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Peripheral blood will be collected from adults ages 18-85. | 2 Years
  These samples will then be used for PCR analysis and T cell cloning.

SECONDARY OUTCOMES:
T cell repertoire | 2 Years
  characterizing the T cell repertoire of individuals with immune mediated skin disease (e.g. psoriasis and mycosis fungoides).

CONTACTS AND LOCATIONS:
Overall Officials: Emanual Maverakis, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical